CLINICAL TRIAL: NCT07030465
Title: Comparison of the Therapeutic Effects of Press Needle and Sham Press Needle on 5-D Pruritus Scale in Hemodialysis Patients With Chronic Kidney Disease-Associated Pruritus
Brief Title: Therapeutic Effects of Press Needle on 5-D Pruritus Scale in Hemodialysis Patients With Chronic Kidney Disease-Associated Pruritus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Visto Pangestu, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 25-06-0788
Record Dates: First submitted 2025-06-12; First posted 2025-06-22 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Chronic Kidney Disease Requiring Chronic Dialysis

STUDY DESIGN:
Intervention Model Description: The press needle, antihistamine, and moisturizer therapy will be designted as the intervention group, while the sham press needle, antihistamine, and moisturizer therapy will be designated as the control group.
Who Masked: Participant, Outcomes Assessor
Masking Description: The participant and outcomes assessor will be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The press needle, antihistamine and moisturizer therapy
  Interventions: Device: The press needle, antihistamine, and moisturizer therapy
- Control Group (Sham Comparator): The sham press needle, antihistamine and moisturizer therapy
  Interventions: Device: The sham press needle, antihistamine and moisturizer therapy

INTERVENTIONS:
Device: The press needle, antihistamine, and moisturizer therapy — Device: Press Needle (PN) PN is applied unilaterally on acupoints LI11, SP10, ST36, and SP6 alternately. It consists of an adhesive patch with a small sterile needle retained for 3-4 days before replacement. This procedure is repeated over a 4-week period. Needle sizes is 0.22 × 1.5 mm), and all procedures follow standard aseptic protocols. PN provides prolonged stimulation with cumulative effects in a minimally invasive manner. Participants continue their routine hemodialysis and conventional treatments for CKD-associated pruritus (CKDaP).
  Arms: Intervention Group
Device: The sham press needle, antihistamine and moisturizer therapy — Sham PN uses adhesive patches without needles, applied to the same acupoints (LI11, SP10, ST36, and SP6) with the same retention schedule (3-4 days over 4 weeks) as the intervention group. All procedures, including placement and instructions, are performed identically to maintain blinding. There is no skin penetration or real acupoint stimulation. Participants continue their routine hemodialysis and conventional treatments for CKDaP.
  Arms: Control Group

SUMMARY:
The goal of this clinical trial is to assess whether press needle acupuncture (PN) is more effective than sham press needle (sham PN) in reducing pruritus in patients with chronic kidney disease-associated pruritus (CKDaP) undergoing hemodialysis. The main questions it aims to answer are:

* Does PN, compared to sham PN, reduce pruritus severity as measured by 5-D Pruritus Scale after the 2nd, 4th, 6th, and 8th therapy sessions?
* Does PN, compared to sham PN, maintain a superior reduction in pruritus severity four weeks after the final session?
* Are there any side effects associated with PN or sham PN in CKDaP patients on hemodialysis?

Participants will:

* Be patients undergoing hemodialysis with confirmed CKDaP
* Undergo cognitive screening with MMSE to ensure accurate self-reporting
* Be randomly assigned to receive either PN (needle inserted) or sham PN (tape only)
* Have PN or sham PN applied unilaterally to acupoints LI11, SP10, ST36, and SP6, replaced every 3-4 days over a 4-week period
* Complete the 5-D Pruritus Scale questionnaire before intervention, after every 2 sessions (2nd, 4th, 6th, 8th), and 4 weeks post-treatment

ELIGIBILITY:
Inclusion Criteria:

* Patients with CKD-associated pruritus (CKDaP) undergoing regular hemodialysis twice a week for at least 6 months and in a hemodynamically stable condition, who meet the criteria for moderate to severe pruritus based on the 5-D Pruritus Scale
* Subjects aged between 18 and 65 years.
* Subjects have not received acupuncture therapy for at least one month prior to the study.
* Subjects have good cognitive function as assessed by the MMSE.
* Subjects are willing to participate in the study according to the scheduled timeline and have signed the informed consent form.

Exclusion Criteria:

* Subjects have malignancies or infectious lesions at the acupuncture points to be treated.
* Subjects have primary skin diseases such as allergic dermatitis, irritant contact dermatitis, neurodermatitis, or psoriasis.
* Subjects have a history of hypersensitivity reactions to previous acupuncture therapy (such as metal allergy, atopy, keloids, or other hypersensitivities).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-10-13 (Actual); Study Completion 2025-10-13 (Actual)

PRIMARY OUTCOMES:
5-D Pruritus Scale | Baseline, after 2nd, 4th, 6th, and 8th treatment sessions, and 4 weeks post-treatment
  Pruritus severity will be assessed using the validated 5-D Pruritus Scale, which evaluates five dimensions: duration, degree, direction, disability, and distribution. Scores range from 5 to 25, with higher scores indicating more severe pruritus.
Adverse events | After 2nd, 4th, 6th, and 8th treatment sessions, and 4 weeks post-treatment
  Any adverse events related to the intervention, including pain, bleeding, skin irritation, or infection at the site of application, will be recorded and monitored.

CONTACTS AND LOCATIONS:
Overall Officials: KPEK FKUI-RSCM, Principal Investigator — The Health Research Ethics Commitee - Faculty of Medicine Universitas Indonesia and Dr. Cipto Mangunkusumo National Hospita
Locations (1):
- Universitas Indonesia, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No